CLINICAL TRIAL: NCT05994950
Title: A Review of the Management and Outcomes of Children With SMA in the West Midlands During 2017-2022
Status: Recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RL1 874
Record Dates: First submitted 2023-07-18; First posted 2023-08-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; Paediatric SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal Muscular Atrophy (SMA) is a rare neuromuscular condition, characterised by loss of motor neurons as a result of a mutation in the survival motor neuron gene. This results in muscle wasting and in the most common and severe type, death before 24 months. Over the recent years there has been a dynamic shift in the therapeutic options for these patients involving both approved therapies, including gene therapy, and access to clinical trials in genetic modifying.

As a result of this mortality and morbidity have changed particularly for the SMA type 1 population and therefore there is now a changing phenotype with many children needing interventions at different time points compared to the natural history. This review process is a retrospective review from 1st July 2017 - 30th June 2022, when most of the new drug therapies were being introduced, of all the children aged from 0-16 years in the West Midlands region and their outcomes.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a rare neuromuscular disorder characterized by degeneration of alpha motor neurons in the spinal cord resulting in progressive muscle wasting, weakness, and paralysis, often leading to early death. It occurs in approximately 1 in 10,000 births. The carrier frequency is variable (between 1:38-1:50) but thought to be highest in Caucasian and Asian populations.

The most common form of SMA is due to a genetic defect in the survival motor neuron 1 (SMN1) gene located on Chromosome 5 (5q11.2-q13.3) which encodes SMN, a protein widely expressed in all eukaryotic cells and necessary for survival of motor neurons. Whilst the diagnosis is made by genetic testing after clinical suspicion, classification is made clinically and on what level of function is achieved, at what age. The severe neonatal type (SMA 0) and the common severe type (SMA I), accounting for approximately 50% cases, presenting before the age of 6 months. These infants, treatment naïve, are very weak and never achieve independent sitting. The rare SMA 0 group generally presents in the neonatal period, often with extreme weakness and contractures and most die within the neonatal period. SMA type II patients present between 6-18 months can achieve independent sitting but are unable to stand and walk and have a reduced life expectancy. SMA type III can be very variable ranging from children who have a similar neuromuscular disability to those with type II, to those that are mildly affected. SMA type IV, the mildest form and very rare, presents in adulthood with onset usually after the second decade, with normal life expectancy. Whilst the sub-groups are classified clinically, there does appear to be a relationship between clinical severity and functional SMN protein and SMN2 copy number. This being said, there has been a phenotypic change since the introduction in the of disease modifying treatment over the last 5 years and therefore the historical classical classification will be evolving. Whilst clinicians have not seen a type I phenotype change to a type II phenotype, many have seen significant changes in mortality and morbidity for these children.

The principle question is how are the West Midlands cohort progressing?

ELIGIBILITY:
Inclusion Criteria:

* Patient aged <16 years old as of 1st July 2017. (16 years old is the age in which patients typically start their transition process to adulthood - retrospective data collection will stop at the date in which the patient turned 16 years old, if this is before 30th June 2022).
* OR patient was born between 1st July 2017 - 30th June 2022.
* Genetically confirmed 5q SMA.
* Patients must have been under the care of the named Key Collaborative Site and Neuromuscular Service for their SMA anytime during 1st July 2017- 30th June 2022 and must have had at least two clinical reviews during this time.
* Deceased patients can be reviewed, as long as they met the eligibility criteria before their date of death.

Exclusion Criteria:

* Aged ≥16 years as of 1st July 2017.
* Genetically confirmed as having non-5q SMA or have no genetic confirmation of their diagnosis.
* Patient was not under the care of the named Key Collaborative Site and Neuromuscular Service for their SMA specialist care anytime during 1st July 2017 - 30th June 2022.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It is important to the methodology of the study that all SMA diagnosed patients known to the services during the timeframe are included in the data collection to evaluate the West Midlands appropriately. The study plans to include a minimum of 30 patients, although the complete patient population known to the service during July 2017- June 2022 that meet the eligibility criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 5 years
  The percentage of patients that passed away between 1st July 2017 - 30th June 2022
Change in Children's Hospital Of Philadelphia Infant Test Of Neuromuscular Disorders (CHOP INTEND) score between 1st July 2017 - 30th June 2022 | 5 years
  Assessing whether the introduction of SMA specific treatment resulted in a change in the CHOP INTEND score over this 5 year period.
Change in Hammersmith Infant Neurological Examination (HINE) score between 1st July 2017 - 30th June 2022 | 5 years
  Assessing whether the introduction of SMA specific treatment resulted in a change in the HINE score over this 5 year period.
Ethnicity | 5 years
  To evaluate whether the patient's ethnicity has an effect on the patient's physical and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Birmingham Heartlands Hospital, Birmingham, Shropshire
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry, Shropshire

IPD SHARING:
Plan to Share IPD: No
The anonymised data set and findings may be reported and disseminated through peer reviewed scientific journals and conference reports. No identifiable data will be used at the time of publication, or throughout the analysis of the data. The anonymised data set may be requested by other researchers with appropriate ethical approval.